CLINICAL TRIAL: NCT06545838
Title: Renin Levels as Prognostic Indicators of Septic Shock Severity and Outcome: Prospective Cohort Study (SOS Trial)
Brief Title: Renin Levels as Prognostic Indicators of Septic Shock Severity and Outcome
Status: Recruiting | Type: Observational
Sponsor: Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Valery Likhvantsev, MD, PhD, Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology
Other Study IDs: SOS
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; Renin; Lactate; Procalcitonin
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic group: Patients with sepsis or septic shock
  Interventions: Other: Analysis of plasma renin concentration

INTERVENTIONS:
Other: Analysis of plasma renin concentration — The concentration of plasma renin in patients will be assessed using the immunochemiluminescent method

SUMMARY:
The Surviving Sepsis Campaign (SSC) of 2021 characterizes sepsis as a life-threatening organ dysfunction caused by a dysregulated host response to infection, with a mortality rate of over 30%, which increases to 40% or more in the case of septic shock. Although concept of sepsis has improved, significant gaps remain in assessing its clinical severity and predicting patient outcomes.

Recognized markers of the severity of septic shock are procalcitonin (PCT), presepsin, and, to a certain extent, lactate. Elevated lactate levels result from a shift to anaerobic glycolysis and indicate inadequate oxygen delivery to tissues. Despite the importance of procalcitonin in the course of sepsis, it has proven to be a suboptimal diagnostic biomarker for the development of sepsis, with sensitivity and specificity below 80%. As a result, the use of procalcitonin in addition to clinical assessment to determine the indications for initiating antibiotic therapy is not recommended. Meanwhile, presepsin, although a potential biomarker for the early diagnosis of sepsis, also has only moderate accuracy according to current data and cannot be used as the only test for the diagnosis of sepsis.

Renin is a crucial enzyme in the renin-angiotensin-aldosterone system (RAAS), which plays an important role in the regulation of blood pressure, tissue perfusion, and the balance of water and electrolytes. Thus, renin may be the sensitive biomarker with good prognostic qualities in the context of sepsis and septic shock. Preliminary studies have indicated that elevated renin levels may act as an indicator of patient severity, and could also be used as a marker for the development of septic shock and mortality prognosis.

This study aims to address these gaps by investigating the role of renin as a biomarker for the severity of sepsis and septic shock, focusing on its potential for more accurate prediction of clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalization in the intensive care unit
* Confirmed diagnosis of Sepsis within 24 hours
* Signed informed consent or a decision by the medical council to include the patient in the study

Exclusion Criteria:

* Any surgical intervention on the kidneys and/or adrenal glands performed within 28 days prior to the patient's inclusion in the study
* Patients previously included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Correlation between blood renin concentration and norepinephrine dosage | Through study completion, an average of 2 years
  A correlation analysis with the calculation of the correlation strength. The degree of correlation ranges from 0 to 1. The closer the correlation coefficient is to one, the stronger the correlation.

SECONDARY OUTCOMES:
Correlation between blood renin concentration and blood procalcitonin concentration | Through study completion, an average of 2 years
  A correlation analysis with the calculation of the correlation strength. The degree of correlation ranges from 0 to 1. The closer the correlation coefficient is to one, the stronger the correlation.
Correlation between blood renin concentration and peripheral blood flow | Through study completion, an average of 2 years
  A correlation analysis with the calculation of the correlation strength. The degree of correlation ranges from 0 to 1. The closer the correlation coefficient is to one, the stronger the correlation.
Correlation between blood renin concentration and SOFA score | Through study completion, an average of 2 years
  A correlation analysis with the calculation of the correlation strength. The degree of correlation ranges from 0 to 1. The closer the correlation coefficient is to one, the stronger the correlation.
Correlation between blood renin concentration and renal replacement therapy free days | Through study completion, an average of 2 years
  A correlation analysis with the calculation of the correlation strength. The degree of correlation ranges from 0 to 1. The closer the correlation coefficient is to one, the stronger the correlation.
28-days mortality | 28 days
  Number of deaths in period of 28 days after enrollment
Frequency of Major Adverse Kidney Events (MAKE) | 28 days
  Count of individuals who experience any of the following: all-cause mortality, renal replacement therapy, and acute kidney injury
Correlation between blood renin concentration and blood lactate concentration | Through study completion, an average of 2 years
  A correlation analysis with the calculation of the correlation strength. The degree of correlation ranges from 0 to 1. The closer the correlation coefficient is to one, the stronger the correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, PhD, Principal Investigator — Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology
Locations (1):
- Federal Research and Clinical Center of Intensive Care Medicine and Rehabilitology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No